CLINICAL TRIAL: NCT05036681
Title: A Phase II Study of Futibatinib and Pembrolizumab in Metastatic Microsatellite Stable Endometrial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0776; NCI-2021-09418 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-08-25; First posted 2021-09-08 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancer; Endometrium Cancer; Endometrial Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Endometrial Neoplasms | interventions — futibatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- futibatini (Experimental)
  Interventions: Drug: Futibatinib
- pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Futibatinib — tablets by mouth 1 time every day
  Arms: futibatini
Drug: Pembrolizumab — Given by vein over about 30-60 minutes on Day 1 of all cycles
  Arms: pembrolizumab

SUMMARY:
It's propose this pilot phase 2 study to explore the combination therapy of futibatinib with pembrolizumab in patients with metastatic microsatellite stable (MSS) endometrial carcinoma to provide a well-tolerated regimen for durable responses.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the objective response rate (ORR) of futibatinib and pembrolizumab in patients with metastatic microsatellite stable (MSS) endometrial carcinoma.
* To evaluate the safety and tolerability.

Primary Endpoints

* Complete responses (CRs) and partial responses (PRs) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Adverse events (AEs: clinical manifestations and laboratory tests) and serious adverse events (SAEs) according to the NCI Common Terminology Criteria for Adverse Events [CTCAE] version 5.0.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this trial, patients must meet all of the following eligibility criteria.

* Patients with histologically confirmed locally advanced or metastatic endometrial carcinoma that is not amenable to curative surgical- or radiation-based intervention, who have received or declined at least one-line systemic chemotherapy.
* Known microsatellite stable (MSS) as pre-identified in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory
* At least one measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Age ≥18 years.
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test prior to administration of the first dose of futibatinib within 7 days prior to initiation of therapy (C1D1), and must agree to use effective birth control initiated immediately following negative serum pregnancy test during screening period, during the study, and for at least 180 days after the last dose (or longer based on local requirements). Female patients are not considered to be of child-bearing potential if they are post-menopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Adequate organ functions as defined below:

Absolute neutrophil count (ANC) ≥ 1,000 /μL. Hemoglobin (Hb) ≥ 9 g/dL. Platelets ≥ 75,000 /μL. Total bilirubin ≤ 1.5 x ULN (upper limit of normal); or total bilirubin < 3 x ULN with direct bilirubin ≤ ULN in patients with well documented Gilbert's Syndrome.

ALT ≤ 3 x ULN or ≤ 5 x ULN if liver metastases persist. Serum phosphate ≤ 1.5 x ULN. Serum calcium ≤ ULN. Serum albumin ≥ 3 g/dL. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance (CrCl) ≥ 40 mL/min by the Cockcroft-Gault method* or 24-hour urine collection.

*CrCl = (140-age) x (weight [kg]) x 0.85 / (72 x serum creatinine mg/dL)

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* No prior treatment with anti-PD-(L)1 therapy and a FGFR inhibitor.
* Ability to read and fully understand the requirements of the trial, willingness to comply with all trial visits and assessments, and willingness and ability to sign an institutional review board (IRB)-approved written informed consent document.
* Any prior radiation must have been completed at least 14 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment (Radiotherapy for extended field within 4 weeks or limited field radiotherapy within 2 weeks).
* Ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may hamper compliance and/or absorption of the study agents (feeding tube is not permitted).
* Provision of an archival tissue block, or 10 formalin-fixed paraffin-embedded (FFPE) slides obtained within 6 months prior to study entry; or agreeing to have biopsies if archival tissues are not available.

Exclusion Criteria:

* Patients who meet any of the following criteria will be not eligible for the study:
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure (New York Heart Association Class III or IV), history of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months before study enrollment, history or current evidence of uncontrolled ventricular arrhythmia. Congenital long QT syndrome, or any known history of torsade de pointes, or family history of unexplained sudden death. Chronic diarrhea diseases considered to be clinically significant in the opinion of the Investigator. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or futibatinib and pembrolizumab administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
* History and/or current evidence of any of the following disorders: Non-tumor related alteration of the calcium-phosphorus homeostasis that is considered clinically significant in the opinion of the Investigator; Ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant in the opinion of the Investigator; and Retinal or corneal disorder confirmed by retinal/corneal examination and considered clinically significant in the opinion of the Investigator and a trained ophthalmologist who performs the test.
* Having not recovered from a major surgical procedure or significant traumatic injury (i.e., still needing additional surgical or medical care for these issues): major surgical procedures ≤ 28 days of treatment entry, or minor surgical procedures ≤ 7 days. No waiting period required following port-a-cath or other central venous access placement.
* Unresolved clinically significant Grade 2 toxicity from prior therapy.
* Patient has an inability to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN).
* Clinically active bleeding, or active gastric or duodenal ulcer.
* Fridericia's corrected QT interval (QTcF =QT/∛(60/HR) ) > 470 ms on ECG conducted during Screening. Patients with an atrioventricular pacemaker or other condition (for example, right bundle branch block) that renders the QT measurement invalid are an exception and the criterion does not apply.
* History of allergic reactions to the study drugs, or any component of the products.
* Currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study. If a patient is currently enrolled in a clinical trial involving non-approved use of a device, then agreement with the investigator and the sponsor is required to establish eligibility.
* Any treatment specifically for systemic tumor control given within 3 weeks before the initiation of the study drugs, within 2 weeks if cytotoxic agents were given weekly, within 6 weeks for nitrosoureas or mitomycin C, within 5 half-lives for targeted agents with half-lives and pharmacodynamic effects lasting < 5 days, or failure to recover from toxic effects of any therapy before the initiation of the study drugs. A drug that has not received regulatory approval for any indication within 14 or 21 days of treatment for a non-myelosuppressive or myelosuppressive agent, respectively.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: Bacille Calmette-Guérin vaccine, measles, mumps, rabies, rubella, typhoid vaccine, varicella/zoster, and yellow fever. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
* Received strong inhibitors and inducers and sensitive substrates of CYP3A4 within 2 weeks (see appendix A).
* Symptomatic primary tumors or metastasis in the brain and/or central nervous system that are uncontrolled with antiepileptics and require steroids at a dose of prednisone > 10 mg/day or equivalent.
* Evidence of leptomeningeal or lymphangitic carcinomatosis.
* A history of another primary malignancy that is currently clinically significant, requiring active intervention except for hormone therapy.
* Concurrent immunosuppressive therapy or steroid (> 10 mg/day prednisone or equivalent).
* Previously documented or suspected autoimmune disease requiring active immunosuppressive therapy (adequately treated skin rash or replacement therapy for endocrinopathies is not excluded), and history of or current pneumonitis.
* Lactation or pregnancy.
* Known human immunodeficiency virus requiring HAART treatment due to unknown drug-drug interactions or known active hepatitis B or C virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siqing fu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one dose level was administered. The trial was terminated due to low enrollment. Enrollment was affected by changes to SOC during the period of trial enrollment
Groups:
- Dose Level 1: Futibatinib 20 mg PO daily Pembrolizumab 200 mg IV on D1
Period: Overall Study
Arm/Group | Dose Level 1
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Objective Response Rate (ORR) of Futibatinib and Pembrolizumab in Patients With Metastatic Microsatellite Stable (MSS) Endometrial Carcinoma.
Time Frame: through study completion, an average of 1 year
Population: Participants were all female, between 50 and 73 of age, all with endometrial cancer
Measure: Number; unit: number of participants with PR/CR
Arm/Group | Dose Level 1
Number analyzed (Participants) | 9
number of participants with PR/CR | 1

ADVERSE EVENTS:
Time Frame: Approximately 2 years 11 months
Arm/Group | Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=9)
Transient ischemic attacl (Nervous system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Generalized weakness (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=9)
Anemia (Blood and lymphatic system disorders) | 5 (15)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (12)
Hyperphosphatemia (Metabolism and nutrition disorders) | 7 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 (4)
Creatinine increased (Investigations) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (3)
White blood cell decreased (Investigations) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify: Hand foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Tumor pain (Eye disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify: elevated prothrombin time (Blood and lymphatic system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycmeia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, specify: COVID-19 infection (Infections and infestations) | 1 (1)
Investigations - Other, specify: decreased total protein (Investigations) | 1 (1)
Investigations - Other, specify: increased TSH (Investigations) | 1 (1)
Keratits (Eye disorders) | 1 (1)
Metabolism and nutritional disorders - Other, specify: elevated serum phosphorus (Metabolism and nutrition disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify: moderate right hydroureteronephrosis (Renal and urinary disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: hard nodules on fingers (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: finger rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: finger warts (Skin and subcutaneous tissue disorders) | 1 (1)
Skin papilloma (Skin and subcutaneous tissue disorders) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ankle frature - Right (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT05036681/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT05036681/ICF_000.pdf